CLINICAL TRIAL: NCT01665430
Title: A Multicenter, Open-Label, Single Arm, Long-Term Extension Study of WA19926 to Describe Safety During Treatment With Tocilizumab in Patients With Early, Moderate to Severe Rheumatoid Arthritis
Brief Title: A Long-Term Extension Study to WA19926 (NCT01007435) of Tocilizumab in Participants With Early, Moderate to Severe Rheumatoid Arthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated by sponsor due to market authorization of tocilizumab for the study population.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28175; 2012-000172-42 (EudraCT Number)
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- Tocilizumab (Experimental): Participants will receive tocilizumab 8 milligrams per kilogram (mg/kg) intravenous infusion every 4 weeks up to 104 weeks.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab will be administered at 8 mg/kg intravenous infusion every 4 weeks, up to 104 weeks.
  Other Names: RoActemra/Actemra

SUMMARY:
This multicenter, open-label, single arm long-term extension of study WA19926 will evaluate the safety and efficacy of tocilizumab (RoActemra/Actemra) in participants with early, moderate to severe rheumatoid arthritis who have completed the WA19926 core study. Eligible participants will receive tocilizumab 8 mg/kg intravenously every 4 weeks for up to 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who complete WA19926 core study (visit at Week 104 and two follow-up telephone visits) and who may benefit from study drug treatment according to the Investigator's assessment
* No current or recent adverse event or laboratory finding preventing the use of the study drug dose of tocilizumab 8 mg/kg at baseline visit
* Receiving treatment on an outpatient basis
* Females of child-bearing potential must agree to use at least one adequate method of contraception as defined by protocol during the treatment period

Exclusion Criteria:

* Pregnant women
* Participants who have prematurely withdrawn from the WA19926 study for any reason
* Treatment with any investigational agent or cell depleting therapies since last administration of study drug in the WA19926 core study
* Treatment with an anti-tumor necrosis factor (TNF) or anti-interleukin (IL)1 agent, or a T-cell co-stimulation modulator since the last administration of the study drug in the WA19926 core study
* Immunization with a live/attenuated vaccine since the last administration of study drug in the WA19926 core study
* Diagnosis since visit at Week 104 of the core WA19926 study of rheumatic autoimmune disease other than rheumatoid arthritis
* Diagnosis since visit at Week 104 of the core WA19926 study of inflammatory joint disease other than rheumatoid arthritis
* Evidence of serious uncontrolled concomitant disease or disorder
* Known active or history of recurrent infection
* Current liver disease as determined by Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Poland (4):
  - Bytom
  - Elblag
  - Poznan
  - Warsaw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included participants with early, moderate to severe rheumatoid arthritis (RA) who had completed WA19926 (NCT01007435) core study and who may have benefited from tocilizumab treatment based on the Investigator's judgment.
Pre-assignment Details: 43 participants were initially screened but only 38 participants were enrolled, and started the study.
Groups:
- Tocilizumab: Participants received tocilizumab 8 milligrams per kilogram (mg/kg) intravenous (IV) infusion every 4 weeks (q4w) up to 104 weeks.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 38
Completed | 29
Not Completed | 9
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 6
Not completed — Other Unspecified | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were enrolled in the study and received at least 1 tocilizumab dose during the study.
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg IV infusion q4w up to 104 weeks.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs), AEs of Special Interest and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs include serious as well as non-serious AEs. AEs of special interest included: Infections including all opportunistic infections and non-serious infections as defined by those treated with IV anti-infectives; Myocardial infarction/acute coronary syndrome; Gastrointestinal perforations and related events; Malignancies; Anaphylaxis/Hypersensitivity reactions; Demyelinating disorders; Stroke; Bleeding events; and Hepatic events.
Time Frame: Baseline up to 112 weeks
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 38
percentage of participants
  AE | 65.8
  AEs of Special Interest | 34.2
  SAE | 7.9

2. Secondary Outcome: Change From Baseline in Disease Activity Index 28 Erythrocyte Sedimentation Rate (DAS28-ESR) Score
Description: DAS28-ESR was calculated from swollen joint count and tender joint count using 28 joints count, erythrocyte sedimentation rate (ESR, in millimeters per hour [mm/hour]) and patient global assessment (PtGA) of disease activity (participant rated arthritis activity assessment on a 0 to 100 millimeter [mm] visual analog scale [VAS]; higher scores indicating greater affectation due to disease activity). Total DAS28-ESR transformed score range: 0 to approximately 10, higher score=more disease activity. Participants who completed the study, or discontinued the study as per sponsor discretion due to marketing authorization approval, were included in End of Study Visit which was Week 104. Participants who withdrew from the study for the reason other than sponsor discretion due to marketing authorization approval, were included in Early Withdrawal Visit. Participants with "Unspecified" reason of discontinuation were excluded for change from baseline analysis.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, at end of study visit (Week 104), at early withdrawal (up to Week 104)
Population: ITT population. Number Analyzed = participants who were evaluable for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 38
units on a scale
  Baseline | 4.365 (1.5502)
  Week 12: number analyzed (Participants) | 35
  Week 12 | -1.832 (1.1985)
  Week 24: number analyzed (Participants) | 34
  Week 24 | -1.496 (1.2683)
  Week 36: number analyzed (Participants) | 31
  Week 36 | -1.904 (1.1682)
  Week 48: number analyzed (Participants) | 32
  Week 48 | -1.970 (1.4503)
  Week 56: number analyzed (Participants) | 32
  Week 56 | -1.979 (1.4368)
  Week 68: number analyzed (Participants) | 30
  Week 68 | -2.069 (1.2486)
  Week 80: number analyzed (Participants) | 24
  Week 80 | -1.831 (1.2592)
  Week 92: number analyzed (Participants) | 13
  Week 92 | -1.792 (1.0792)
  End of Study: number analyzed (Participants) | 29
  End of Study | -2.187 (1.1785)
  Early Withdrawal: number analyzed (Participants) | 7
  Early Withdrawal | -1.624 (1.8930)

3. Secondary Outcome: Change From Baseline in Total Tender Joint Counts (28 Joints)
Description: The number of tender joints was recorded on the joint assessment form, no tenderness = 0, tenderness = 1, for 28 joints and joints were classified as tender/not tender giving a total possible tender joint count of 0 to 28. Participants who completed the study, or discontinued the study as per sponsor discretion due to marketing authorization approval, were included in End of Study Visit which was Week 104. Participants who withdrew from the study for the reason other than sponsor discretion due to marketing authorization approval, were included in Early Withdrawal Visit. Participants with "Unspecified" reason of discontinuation were excluded for change from baseline analysis.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, at end of study visit (Week 104), at early withdrawal (up to Week 104)
Population: ITT population. Number Analyzed = participants who were evaluable for specified category.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 38
tender joints
  Baseline | 12.6 (16.54)
  Week 12: number analyzed (Participants) | 35
  Week 12 | -7.7 (12.63)
  Week 24: number analyzed (Participants) | 34
  Week 24 | -5.0 (10.95)
  Week 36: number analyzed (Participants) | 32
  Week 36 | -6.1 (13.13)
  Week 48: number analyzed (Participants) | 32
  Week 48 | -6.1 (11.17)
  Week 56: number analyzed (Participants) | 32
  Week 56 | -7.6 (11.89)
  Week 68: number analyzed (Participants) | 30
  Week 68 | -7.2 (9.63)
  Week 80: number analyzed (Participants) | 24
  Week 80 | -10.0 (13.74)
  Week 92: number analyzed (Participants) | 13
  Week 92 | -6.9 (16.10)
  End of Study: number analyzed (Participants) | 29
  End of Study | -9.3 (13.61)
  Early Withdrawal: number analyzed (Participants) | 7
  Early Withdrawal | -6.1 (9.51)

4. Secondary Outcome: Change From Baseline in Total Swollen Joint Counts (28 Joints)
Description: The number of swollen joints was recorded on the joint assessment form, no swelling = 0, swelling =1, for 28 joints and were classified as swollen/not swollen giving a total possible swollen joint count of 0 to 28. Participants who completed the study, or discontinued the study as per sponsor discretion due to marketing authorization approval, were included in End of Study Visit which was Week 104. Participants who withdrew from the study for the reason other than sponsor discretion due to marketing authorization approval, were included in Early Withdrawal Visit. Participants with "Unspecified" reason of discontinuation were excluded for change from baseline analysis.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, at end of study visit (Week 104), at early withdrawal (up to Week 104)
Population: ITT population. Number Analyzed = participants who were evaluable for specified category.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 38
swollen joints
  Baseline | 4.8 (4.67)
  Week 12: number analyzed (Participants) | 35
  Week 12 | -2.5 (3.42)
  Week 24: number analyzed (Participants) | 34
  Week 24 | -2.0 (3.24)
  Week 36: number analyzed (Participants) | 32
  Week 36 | -2.1 (3.61)
  Week 48: number analyzed (Participants) | 32
  Week 48 | -2.4 (3.90)
  Week 56: number analyzed (Participants) | 32
  Week 56 | -2.7 (3.91)
  Week 68: number analyzed (Participants) | 30
  Week 68 | -2.9 (3.90)
  Week 80: number analyzed (Participants) | 24
  Week 80 | -2.5 (4.42)
  Week 92: number analyzed (Participants) | 13
  Week 92 | -3.0 (5.45)
  End of Study: number analyzed (Participants) | 29
  End of Study | -2.8 (4.12)
  Early Withdrawal: number analyzed (Participants) | 7
  Early Withdrawal | -4.3 (5.28)

5. Secondary Outcome: Percentage of Participants With Drug-Free Remission
Description: Drug-free remission was defined as having clinical remission (defined as DAS28-ESR score <2.6) for 2 consecutive assessment visits followed by discontinuation of tocilizumab at the second assessment visit. DAS28-ESR was calculated from swollen joint count and tender joint count using 28 joints count, ESR, (mm/hour) and PtGA of disease activity (participant rated arthritis activity assessment on a 0 to 100 mm VAS; higher scores indicating greater affectation due to disease activity). Total DAS28-ESR transformed score range: 0 to approximately 10, higher score=more disease activity.
Time Frame: Baseline up to Week 104 (assessed at Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, at end of study visit [Week 104], at early withdrawal [up to 104 weeks])
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 38
percentage of participants | 0.0

6. Secondary Outcome: Percentage of Participants With Clinical Remission
Description: Clinical remission was defined as having DAS28-ESR score <2.6 at any point during the study. DAS28-ESR was calculated from swollen joint count and tender joint count using 28 joints count, ESR, (mm/hour) and PtGA of disease activity (participant rated arthritis activity assessment on a 0 to 100 mm VAS; higher scores indicating greater affectation due to disease activity). Total DAS28-ESR transformed score range: 0 to approximately 10, higher score=more disease activity.
Time Frame: as for outcome 5
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 38
percentage of participants | 81.6

7. Secondary Outcome: Time to Rheumatoid Arthritis (RA) Flare in Participants Who Had Entered Drug-Free Remission
Description: Time to RA flare was defined as the period of drug-free remission (having DAS28-ESR score <2.6 for 2 consecutive assessment visits followed by discontinuation of tocilizumab at the second assessment visit) until documented RA flare. RA flare was defined as any worsening of the participant's disease activity that, in the opinion of the Investigator, required treatment intensification beyond supportive therapy which could include restarting the study drug.
Time Frame: as for outcome 5
Population: The time to RA flare could not be evaluated as none of the participants showed drug-free remission.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Physician's Global Assessment (PGA) of Disease Activity Using Visual Analog Scale (VAS)
Description: The PGA of disease activity was assessed using a 0 to 100 mm horizontal VAS by the physician. The left-hand extreme of the line equaled 0 mm, and was described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equaled 100 mm, and was described as "maximum disease activity" (maximum arthritis disease activity). A negative change from baseline indicated improvement. Participants who completed the study, or discontinued the study as per sponsor discretion due to marketing authorization approval, were included in End of Study Visit which was Week 104. Participants who withdrew from the study for the reason other than sponsor discretion due to marketing authorization approval, were included in Early Withdrawal Visit. Participants with "Unspecified" reason of discontinuation were excluded for change from baseline analysis.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, at end of study visit (Week 104), at early withdrawal (up to 104 weeks)
Population: ITT population. Number Analyzed = participants who were evaluable for specified category.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 38
mm
  Baseline | 32.1 (24.60)
  Week 12: number analyzed (Participants) | 35
  Week 12 | -15.1 (21.57)
  Week 24: number analyzed (Participants) | 34
  Week 24 | -16.0 (19.05)
  Week 36: number analyzed (Participants) | 32
  Week 36 | -17.3 (19.37)
  Week 48: number analyzed (Participants) | 32
  Week 48 | -18.0 (20.06)
  Week 56: number analyzed (Participants) | 32
  Week 56 | -19.0 (20.60)
  Week 68: number analyzed (Participants) | 30
  Week 68 | -20.6 (22.13)
  Week 80: number analyzed (Participants) | 24
  Week 80 | -19.2 (19.01)
  Week 92: number analyzed (Participants) | 13
  Week 92 | -21.2 (17.50)
  End of Study: number analyzed (Participants) | 29
  End of Study | -22.2 (20.92)
  Early Withdrawal: number analyzed (Participants) | 7
  Early Withdrawal | -2.9 (22.71)

9. Secondary Outcome: Change From Baseline in PtGA of Disease Activity Using VAS
Description: The PtGA of disease activity was assessed using a 0 to 100 mm horizontal VAS by the participant. The left-hand extreme of the line equaled 0 mm, and was described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equaled 100 mm, and was described as "maximum disease activity" (maximum arthritis disease activity). A negative change from baseline indicated improvement. Participants who completed the study, or discontinued the study as per sponsor discretion due to marketing authorization approval, were included in End of Study Visit which was Week 104. Participants who withdrew from the study for the reason other than sponsor discretion due to marketing authorization approval, were included in Early Withdrawal Visit. Participants with "Unspecified" reason of discontinuation were excluded for change from baseline analysis.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, at end of study visit (Week 104), at early withdrawal (up to 104 weeks)
Population: ITT population. Number Analyzed = participants who were evaluable for specified category.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 38
mm
  Baseline | 34.9 (27.33)
  Week 12: number analyzed (Participants) | 35
  Week 12 | -10.1 (21.63)
  Week 24: number analyzed (Participants) | 34
  Week 24 | -6.4 (20.57)
  Week 36: number analyzed (Participants) | 32
  Week 36 | -11.4 (20.14)
  Week 48: number analyzed (Participants) | 32
  Week 48 | -9.1 (21.24)
  Week 56: number analyzed (Participants) | 32
  Week 56 | -8.5 (19.14)
  Week 68: number analyzed (Participants) | 30
  Week 68 | -11.0 (21.54)
  Week 80: number analyzed (Participants) | 24
  Week 80 | -16.0 (24.10)
  Week 92: number analyzed (Participants) | 13
  Week 92 | -12.8 (12.40)
  End of Study: number analyzed (Participants) | 29
  End of Study | -16.4 (22.13)
  Early Withdrawal: number analyzed (Participants) | 7
  Early Withdrawal | 5.4 (34.88)

10. Secondary Outcome: Change From Baseline in Participant Assessment of Pain Using VAS
Description: Severity of pain was evaluated by a VAS. Participants marked on a 100 mm horizontal VAS the severity of pain that they had experienced because of their RA, ranging from 0 mm (no pain) to 100 mm (unbearable pain). Participants who completed the study, or discontinued the study as per sponsor discretion due to marketing authorization approval, were included in End of Study Visit which was Week 104. Participants who withdrew from the study for the reason other than sponsor discretion due to marketing authorization approval, were included in Early Withdrawal Visit. Participants with "Unspecified" reason of discontinuation were excluded for change from baseline analysis.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, at end of study visit (Week 104), at early withdrawal (up to 104 weeks)
Population: ITT population. Number Analyzed = participants who were evaluable for specified category.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 38
mm
  Baseline | 35.0 (26.48)
  Week 12: number analyzed (Participants) | 35
  Week 12 | -11.6 (20.80)
  Week 24: number analyzed (Participants) | 34
  Week 24 | -8.4 (19.74)
  Week 36: number analyzed (Participants) | 32
  Week 36 | -12.7 (19.05)
  Week 48: number analyzed (Participants) | 32
  Week 48 | -10.9 (19.96)
  Week 56: number analyzed (Participants) | 32
  Week 56 | -9.9 (19.71)
  Week 68: number analyzed (Participants) | 30
  Week 68 | -11.7 (20.16)
  Week 80: number analyzed (Participants) | 24
  Week 80 | -15.3 (22.22)
  Week 92: number analyzed (Participants) | 13
  Week 92 | -10.9 (13.59)
  End of Study: number analyzed (Participants) | 29
  End of Study | -17.2 (20.13)
  Early Withdrawal: number analyzed (Participants) | 7
  Early Withdrawal | -0.7 (32.62)

11. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The HAQ-DI was a participant self-reported questionnaire for assessing the extent of a participant's functional ability. It consisted of 20 questions in 8 categories (dressing and grooming, rising, eating, walking, reach, grip, hygiene, and carrying out daily activities). Each question had 4 response options, ranging from 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. The HAQ-DI scale was an average of all the scores from all questions and ranged from 0 to 3, where higher scores represented higher disease activity. Participants who completed the study, or discontinued the study as per sponsor discretion due to marketing authorization approval, were included in End of Study Visit which was Week 104. Participants who withdrew from study for reason other than sponsor discretion due to marketing authorization approval, were included in Early Withdrawal Visit. Participants with "Unspecified" reason of discontinuation were excluded for change from baseline analysis.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, at end of study visit (Week 104), at early withdrawal (up to 104 weeks)
Population: ITT population. Number Analyzed = participants who were evaluable for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 38
units on a scale
  Baseline | 0.871 (0.5981)
  Week 12: number analyzed (Participants) | 35
  Week 12 | -0.169 (0.3255)
  Week 24: number analyzed (Participants) | 34
  Week 24 | -0.163 (0.4301)
  Week 36: number analyzed (Participants) | 32
  Week 36 | -0.208 (0.4965)
  Week 48: number analyzed (Participants) | 32
  Week 48 | -0.106 (0.5001)
  Week 56: number analyzed (Participants) | 32
  Week 56 | -0.185 (0.5024)
  Week 68: number analyzed (Participants) | 30
  Week 68 | -0.076 (0.4154)
  Week 80: number analyzed (Participants) | 24
  Week 80 | -0.152 (0.4095)
  Week 92: number analyzed (Participants) | 13
  Week 92 | -0.271 (0.3100)
  End of Study: number analyzed (Participants) | 29
  End of Study | -0.239 (0.5698)
  Early Withdrawal: number analyzed (Participants) | 7
  Early Withdrawal | 0.019 (0.2230)

ADVERSE EVENTS:
Time Frame: Baseline up to 112 weeks
Description: ITT population.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 3/38
Other Adverse Events (participants affected / at risk) | 22/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=38)
Vestibular neuronitis (Infections and infestations) | 1
Myocardial ischemia (Cardiac disorders) | 1
Speech disorder (Nervous system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=38)
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 4
Bronchitis (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 11
Hepatic enzyme increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6
Dyslipidaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2

LIMITATIONS AND CAVEATS:
The study was terminated due to sponsor decision which was due to market authorization of tocilizumab for the treatment of severe, active and progressive RA in adults not previously treated with methotrexate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.